CLINICAL TRIAL: NCT03242928
Title: A Randomized, Subject and Investigator Blinded, Placebo-controlled, Parallel Group Study to Investigate Whether AFQ056 Reduces Cocaine Use in Patients Diagnosed With Cocaine Use Disorder (CUD)
Brief Title: Study to Investigate Whether AFQ056 Reduces Cocaine Use in Patients Diagnosed With Cocaine Use Disorder (CUD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAFQ056X2201; 2017-000736-33 (EudraCT Number)
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Results first posted 2021-02-04 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Cocaine-related Disorder
Keywords: Cocaine Use Disorder; cocaine dependence,AFQ056,adult, cocaine use,CUD, drug abuse, drug addiction,
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matching tablet of placebo taken orally BID
  Interventions: Drug: Placebo
- AFQ056 (Experimental): Mavoglurant was up titrated on a bid regimen followed by fixed-dose bid regimen: 50 mg bid from Day 1 to Day 7, 100 mg bid from Day 8 to Day 14, and then fixed-dose 200 mg bid for 84 days
  Interventions: Drug: AFQ056

INTERVENTIONS:
Drug: AFQ056 — 50 mg and 100 mg tablets taken orally
  Other Names: mavoglurant
  Arms: AFQ056
Drug: Placebo — Matching placebo tablets taken orally BID
  Arms: Placebo

SUMMARY:
This study assessed whether AFQ056 had a beneficial effect by reducing cocaine use in Cocaine Use Disorder (CUD) patients as assessed by Timeline Follow-Back cocaine self-report.

DETAILED DESCRIPTION:
This was a randomized, subject- and Investigator-blinded, parallel-group, placebo-controlled study in subjects with CUD. The study consisted of a 17-day screening period followed by a 12-day baseline, a 98-day outpatient treatment period (14-day up-titration dose regimen followed by 84-day maintenance dose), and an End of Study evaluation visit approximately 14 days after the last study drug administration. The total duration for each subject in the study was approximately 20 weeks including screening and baseline.

ELIGIBILITY:
Inclusion Criteria:

* Understand the study procedures and provide written informed consent before any assessment is performed.
* Subjects diagnosed with Cocaine Use Disorder according to DSM 5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Ed.).
* Must use cocaine through snorting (intranasally) as primary route of administration.
* Recent cocaine use confirmed by positive urine screen for 1 or more benzoylecgonine (BE).
* Must be seeking treatment for cocaine dependence and have a desire to reduce or cease cocaine use.

Exclusion Criteria:

* Has current diagnosis of Substance Use Disorder (according to the DSM 5) on alcohol, cannabis or other stimulants, except cocaine.
* Meets current or lifetime DSM 5 criteria for schizophrenia or any psychotic disorder, or organic mental disorder.
* Have current treatment for Substance Use Disorder (e.g.: disulfiram, acamprosate, methyl phenidate, modafinil, topiramate, immediate release dexamfetamine,or baclofen).
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
* Have a history of any illness, condition, and use of medications that in the opinion of the investigator or designee might confound the results of the study or pose additional risk in administering the investigational agents to the subject or preclude successful completion of the study
* Current or/and previous treatment with concomitant medications that are strong or moderate inducers/inhibitors of CYP3A4 (e.g., clarithromycin, ketoconazole, ritonavir, etc.)
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
* Chronic infection with Hepatitis B (HBV) or Hepatitis C (HCV).
* Score "yes" on item 4 or item 5 of the Suicidal Ideation section of the CSSRS, if this ideation occurred in the past 6 months, or "yes" on any item of the Suicidal Behavior section, except for the "Non-Suicidal Self-Injurious Behavior" (item also included in the Suicidal Behavior section), if this behavior occurred in the past 2 years.
* Controlled hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Novartis Investigative Site, Buenos Aires, Argentina
- Spain (3):
  - Novartis Investigative Site, Sant Joan d'Alacant, Alicante
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Zurich

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to to respect the privacy of patients who have participated in the trail in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalsutdydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=689

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 68 patients who received study treatment.
Period: Overall Study
Arm/Group | AFQ056 | Placebo
Started | 31 | 37
Completed | 22 | 32
Not Completed | 9 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AFQ056 | Placebo | Total
Number analyzed (Participants) | 31 | 37 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (8.31) | 35.5 (9.19) | 35.4 (8.74)
Age, Customized [Number; unit: Participants]
  18 - 65 years | 31 | 37 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 26 | 30 | 56
Race/Ethnicity, Customized [Number; unit: participants]
  White | 31 | 36 | 67
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Cocaine Use Days
Description: The cocaine consumption was recorded once daily (Yes/No) by the subject using the Timeline Follow-Back (TLFB) cocaine assessment tool during the treatment period. For each patient, the proportion of cocaine use days was calculated by dividing the number of days of cocaine use during the treatment period, i.e. 98 days for completers and number of days between Day 1 and day of last dose in case of premature discontinuation of study treatment.
Time Frame: Day 1 up to day 98
Population: Pharmacodynamic analysis set (PD): subjects with any available efficacy (PD) data, who received study drug for at least 14 days with no relevant protocol deviation
Measure: Mean (Standard Error); unit: cocaine use days
Arm/Group | AFQ056 | Placebo
Number analyzed (Participants) | 29 | 36
cocaine use days | 0.122 (0.027) | 0.209 (0.024)
Statistical Analysis 1: Comparison: AFQ056 vs Placebo; Test type: Superiority; p = 0.021, ANCOVA; Mean Difference (Final Values) = -0.087, 95% CI 2-sided [-0.161 to -0.013], Standard Error of Mean 0.037

2. Secondary Outcome: Proportion of Positive Urine Measurements of Benzoylecgonine (BE)
Description: Urine samples were analyzed for the presence of cocaine's metabolite benzoylecgonine (BE) which is the main metabolite of cocaine present in urine. Two urine samples were provided per week to provide a quantitative measure.
Time Frame: Day 1 up to day 98
Measure: Mean (Standard Error); unit: positive urine samples
Arm/Group | AFQ056 | Placebo
Number analyzed (Participants) | 29 | 36
positive urine samples | 0.666 (0.057) | 0.843 (0.051)
Statistical Analysis 1: Comparison: AFQ056 vs Placebo; Test type: Superiority; p = 0.025, ANOVA; Mean Difference (Final Values) = -0.177, 95% CI 2-sided [-0.331 to -0.023], Standard Error of Mean 0.077

3. Secondary Outcome: Proportion of Days of Alcohol Consumption
Description: Alcohol consumption was recorded by the subjects using the Timeline Follow-Back (TLFB) alcohol self report. The number of standard drinks were recorded daily. The proportion of days of alcohol consumption during the study treatment period was was compared using an ANCOVA model with treatment as factor and past alcohol consumption as covariate. The past consumption of alcohol was the proportion of alcohol over the 28 days preceding the screening visit, which was assessed retrospectively using the TLFB.
Time Frame: Day 1 up to day 98
Population: as for outcome 1
Measure: Mean (Standard Error); unit: alcohol consumption days
Arm/Group | AFQ056 | Placebo
Number analyzed (Participants) | 29 | 36
alcohol consumption days | 0.233 (0.030) | 0.303 (0.026)
Statistical Analysis 1: Comparison: AFQ056 vs Placebo; Test type: Superiority; p = 0.072, ANCOVA; Mean Difference (Final Values) = -0.070, 95% CI 2-sided [-0.146 to 0.006], Standard Error of Mean 0.038

4. Secondary Outcome: AFQ056 Plasma Concentrations
Description: Plasma samples were collected to assess pharmacokinetics (PK)
Time Frame: Day 15 (0h, 2h), Day 29 (0, 2h), Day 57 (0h, 2h), Day 98 (0h,2h)
Population: Number of samples available for analysis varied across time points
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AFQ056
Number analyzed (Participants) | 29
ng/mL
  Day 15 0 hour: number analyzed (Participants) | 21
  Day 15 0 hour | 41.2 (47.4)
  Day 15 2 hour: number analyzed (Participants) | 21
  Day 15 2 hour | 78.0 (91.7)
  Day 29 0 hour: number analyzed (Participants) | 26
  Day 29 0 hour | 83.5 (116)
  Day 29 2 hour: number analyzed (Participants) | 24
  Day 29 2 hour | 148 (131)
  Day 57 0 hour: number analyzed (Participants) | 22
  Day 57 0 hour | 108 (153)
  Day 57 2 hour: number analyzed (Participants) | 22
  Day 57 2 hour | 141 (153)
  Day 98 0 hour: number analyzed (Participants) | 21
  Day 98 0 hour | 89.8 (148)
  Day 98 2 hour: number analyzed (Participants) | 21
  Day 98 2 hour | 116 (86.1)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 14 days post treatment, up to maximum duration of approximately 16 weeks
Arm/Group | AFQ056 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/31 | 1/37
Other Adverse Events (participants affected / at risk) | 26/31 | 30/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AFQ056 (N=31) | Placebo (N=37)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AFQ056 (N=31) | Placebo (N=37)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 3 (3) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (6) | 7 (12)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 2 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (8) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 6 (6)
Vomiting (Gastrointestinal disorders) | 3 (6) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (4) | 3 (3)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (4) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Physical deconditioning (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Thirst (General disorders) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 4 (7) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 8 (10)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (3)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine abnormal (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 3 (3) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (2)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Red blood cell count increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (6)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 7 (17) | 4 (4)
Headache (Nervous system disorders) | 6 (13) | 10 (24)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (3) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Resting tremor (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 4 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (4) | 4 (5)
Aversion (Psychiatric disorders) | 1 (3) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 2 (3)
Depression (Psychiatric disorders) | 1 (3) | 0 (0)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (2)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0)
Feeling guilty (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, olfactory (Psychiatric disorders) | 1 (3) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 2 (3) | 0 (0)
Ideas of reference (Psychiatric disorders) | 0 (0) | 2 (2)
Illusion (Psychiatric disorders) | 2 (2) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (9) | 2 (11)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2)
Nightmare (Psychiatric disorders) | 2 (2) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 3 (4) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal mucosal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (7) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03242928/Prot_001.pdf
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT03242928/SAP_000.pdf